CLINICAL TRIAL: NCT06346873
Title: Pilot Study to Demonstrate Efficacy of JOGO for the Treatment of Tremor
Brief Title: Demonstrating Efficacy of JOGO for the Treatment of Tremor
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI No longer at Mayo Clinic
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-008090
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Functional Neurological Disorder
Keywords: Functional Tremor
MeSH Terms: conditions — Conversion Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- JOGO for the Treatment of Tremor (Experimental): Subjects with a diagnosis of essential tremor (ET) or functional tremor (FT) involving one or more of the upper extremities will undergo a 12-week JOGO treatment program.
  Interventions: Device: JOGO

INTERVENTIONS:
Device: JOGO — AI driven mobile app and wearable sensors to provide virtual treatments

SUMMARY:
This research is being done to determine the effectiveness of a new treatment, called JOGO, for patients with functional tremor (FT). JOGO is a biofeedback device that has been shown to help patients with several conditions, e.g., chronic pain, migraine, and Parkinson's disease (PD)-related tremor. JOGO provides biofeedback by using wireless adhesive stickers, called surface electromyography, to get information about muscle activity. This information is then used to modify symptoms through a series of training sessions with a physical therapist and individual practice.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of functional tremor diagnosed by a Mayo Clinic Florida movement disorders specialist.
* Must have access to reliable internet video.

Exclusion Criteria:

* Cognitive impairment (Montreal Cognitive Assessment greater than 26).
* Currently taking any of the following medications to treat tremor: primidone, gabapentin, zonisamide, any non-selective beta blocker, any benzodiazepine.
* Exposure to tremorgenic drugs or drug with withdrawal states within 30 days prior to the study start.
* Direct or indirect trauma to the nervous system within 3 months preceding the onset of tremor.
* Known history of other medical or neurological conditions that may cause or explain subject's tremor, including, but not limited to: Parkinson's disease, dystonia, cerebellar disease, traumatic brain injury, alcohol abuse or withdrawal, mercury poisoning, hyperthyroidism, pheochromocytoma, head trauma or cerebrovascular disease within 3 months prior to the onset of essential tremor, multiple sclerosis, polyneuropathy, family history of Fragile X syndrome.
* Prior MR-guided focused ultrasound or surgical intervention (e.g., deep brain stimulation, ablative thalamotomy or gamma knife thalamotomy).
* Botulinum toxin injection in the 6 months prior to screening.
* Use of medication(s) in the past month that might produce tremor or interfere with the evaluation of tremor, such as, but not limited to: CNS-stimulants, lithium, amiodarone, metoclopramide, theophylline, and valproate.
* Regular use of more than two units of alcohol per day.
* Sporadic use of a benzodiazepine, sleep medication or anxiolytic to improve sleep performance. Stable use at a consistent dose is allowed if tremor persists against the background of regular medication use.
* Current treatment with any investigational therapy for tremor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-03 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-01-03 (Actual)

PRIMARY OUTCOMES:
Change in TETRAS scores 1 month | Baseline, 1-month post-treatment
  Assessment with The Essential Tremor Rating Assessment Scale (TETRAS), consists of ten items in which action tremor is rated 0-4 in half-point increments by a clinician. Greater total scores indicate worse action tremor.

SECONDARY OUTCOMES:
Change in TETRAS scores 2 months | Baseline, 2-month post-treatment
  Assessment with The Essential Tremor Rating Assessment Scale (TETRAS), consists of ten items in which action tremor is rated 0-4 in half-point increments by a clinician. Greater total scores indicate worse action tremor.
Change in QUEST scores | Baseline, 1-month and 2-month post-treatment
  Measured by self-assessment with the Quality of Life in Essential Tremor Questionnaire (QUEST)
Tremor prevalence | 2 months
  Number of tremors in time awake during the day measured by wearable device system (KinesiaUTM).
Tremor resolution 1 month | 1-month post-treatment
  Number of subjects to experience tremor resolution on in-lab assessment
Tremor resolution 2 months | 2-months post-treatment
  Number of subjects to experience tremor resolution on in-lab assessment
Change in BDI-II scores | Baseline, 1-month and 2-month post-treatment
  Assessment with the Beck Depression Index II (BDI-II) questionnaire to assess depression severity, a 21-item scale, with items ranging from 0 to 3. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.
Change in BAI scores | Baseline, 1-month and 2-month post-treatment
  Assessment with the Beck Anxiety Index (BAI) that measures the severity of anxiety symptoms. Possible scores range from 0 to 63 with higher scores indicating a worse outcome/more severe symptoms of anxiety.
Change in Intolerance of Uncertainty Scale | Baseline, 1-month and 2-month post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Philip Tipton, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials